CLINICAL TRIAL: NCT04181047
Title: RCT Investigating Virtual Eye Movement Desensitization and Reprocessing (EMDR) for Adults With Suicidal Ideation
Brief Title: RCT Investigating EMDR for Suicidal Ideation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090989
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Suicidal Ideation
Keywords: Eye movement desensitization and Reprocessing, Suicide
MeSH Terms: conditions — Suicidal Ideation; Suicide | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Non-blinded randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual EMDR (Experimental): Patients will receive 1 to 3 preparation sessions (which will include psychoeducation and preparation exercises before EMDR), followed by up to 12 EMDR sessions, delivered over encrypted Zoom videoconferencing. EMDR is an evidence based trauma therapy. These EMDR sessions will focus on the experiences, urges or negative thoughts associated with their suicidal thoughts. The sessions will be 90 minutes in length and occur twice per week. This group will also have access to usual psychiatric care, which usually includes a family doctor or psychiatrist, mental health therapist and having access to Edmonton's community mental health programs.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR); Other: Usual care
- Treatment as usual (Active Comparator): This group will also have access to usual care, which usually includes a family doctor or psychiatrist, mental health therapist and having access to Edmonton's community mental health programs.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — Psychotherapy.
  Arms: Virtual EMDR
Other: Usual care — Access to usual care, including psychiatrist, medications, mental health therapist, general community mental health programs. TAU will NOT include electroconvulsive therapy or another trauma specific psychotherapy.

SUMMARY:
Suicide is a major public health issue, and is the 9th leading cause of death overall. Suicidal thinking and behaviours have been linked to painful childhood experiences, stressors, and psychological trauma. Stressful experiences are also strongly linked to the development of a variety of mental health problems, including anxiety, depression and posttraumatic stress disorder. However, patients with suicidal ideas are often left out of trauma treatment, for fear that it will worsen their distress and increase their suicidal thinking. However, there is preliminary evidence that treating posttraumatic stress symptoms in patients with suicidal thoughts can lead to improvement in their symptoms and a reduction in suicidal thinking.

For many individuals, overwhelming emotions and/or painful negative beliefs stemming from traumatic experiences contribute to a desire to escape though suicide or self-harm. Eye Movement Desensitization and Reprocessing (EMDR) is an evidence-based therapy for posttraumatic stress disorder that desensitizes painful memories, so that reminders in the present no longer provoke the overwhelming emotional responses. It has also been used for depression and a variety of other mental health problems.

This study aims to test the safety and effectiveness of virtual/remotely delivered EMDR for adults with suicidal ideation. Patients will be randomly assigned to receive either EMDR therapy plus Treatment as usual (TAU) or TAU alone. Symptoms of anxiety, depression, post-traumatic stress, distressing emotions, and suicidal thinking will be compared before and after therapy. For the EMDR group, side effects to EMDR will be tracked. The number of emergency room visits and hospitalizations will also be compared before and after therapy for each group.

DETAILED DESCRIPTION:
Suicide is the second leading cause of death among those aged 10-29 years, the 9th leading cause of death overall, and there are 4000 completed suicides per year in Canada. Adverse childhood experiences, interpersonal stressors and trauma correlate strongly with suicidal behaviour and the later development of psychopathology such as depression. For many individuals, overwhelming emotions and/or painful negative beliefs stemming from traumatic experiences contribute to a desire to escape though suicide or self-harm. Eye Movement Desensitization and Reprocessing (EMDR) is an evidence-based therapy for posttraumatic stress disorder that desensitizes painful memories, so that reminders in the present no longer provoke the overwhelming emotional responses.

The COVID-19 pandemic has forced a rapid shift from in-person psychotherapy to remotely delivered psychotherapy services, both to reduce the spread of COVID-19 as well as to maintain access to services. Given this rapid shift to remote delivery and the need for a review of evidence, a recent systematic scoping review was undertaken regarding the scope and quality of peer reviewed literature on remotely delivered psychotherapeutic digital health interventions for military members, veterans and public safety personnel with posttraumatic stress injury (Jones et al 2020). This review yielded 38 studies for inclusion, demonstrating level 1a evidence for prolonged exposure therapy, cognitive processing therapy, behavioral activation and therapeutic exposure in this population. There was evidence that remote delivery of these therapies can be as effective as in-person treatment, and also possibly reduce stigma and improve access to care. There was limited information about EMDR, despite the fact that online EMDR has been widely adopted around the world clinically.

This project had originally aimed to enroll inpatients in face to face therapy and transition them to the outpatient environment. However, the COVID-19 pandemic has resulted in shorter inpatient length of stay, extremely limited mobility for inpatients on and off the units, and shortages of appropriate spaces, making this untenable. There has also been an increase in demand for mental health services at the same time as a reduction in availability of in-person mental health supports. Furthermore, public health measures have necessitated periodic self-isolation, leading to clinic cancellations. For all these reasons, this project will deliver EMDR via Zoom videoconferencing, rather than in person.

This real-world, non-blinded randomized study aims to evaluate the safety and efficacy of EMDR for adults (ages 18 to 65) with suicidal ideation. Eighty participants will be randomized into one of two groups. Group one will receive EMDR therapy to desensitize and reprocess the experiences associated with suicidal thinking. This will be delivered online via encrypted Zoom, due to the COVID-19 pandemic. Group two will be randomized to "treatment as usual" (TAU), which will serve as a control group. TAU will include regular psychiatric care. Clinical measures of anxiety, depression, post-traumatic symptoms, emotional dysregulation, and suicidal thinking will be compared before and after therapy. The impact on emergency room visits, re-hospitalizations and healthcare costs will also be evaluated one year after study completion.

ELIGIBILITY:
Inclusion criteria include

1. adults (ages 18 to 65) with suicidal ideation in the last week.
2. Participants must volunteer to be in the study, be able to give informed consent and be able to follow up twice weekly until treatment is complete (a total of 12 sessions).
3. Participants must have a primary service provider.
4. Participants must have access to their own laptop or desktop computer that enables BLS with a working screen, camera, and microphone, and access to a quiet, private, well-lit space for therapy.
5. Participants must be willing to refrain from benzodiazepine, cannabis or illicit substance use in the 24 hours before or after EMDR sessions.
6. Participants must be willing to adhere to the study safety precautions

Exclusion criteria

1. At the time of assessment, suicidal ideation is not accompanied by intent or plan to follow through with suicide.
2. Known pregnancy, as there is limited information about the impact of EMDR in pregnancy.
3. DES score above 34 or severe dissociative symptoms (see below), psychotic symptoms or manic symptoms.
4. Participants undergoing or planning to undergo electroconvulsive therapy (ECT) or another trauma focused psychotherapy in the 4-month study period.

Referred potential participants will also be excluded on the basis of the assessment interview if they report a history of severe dissociative symptoms in keeping with a separate dissociative disorder, such as

1. hearing internal voices,
2. amnestic episodes, or dissociative fugue states
3. passivity experiences or first rank symptoms under stress, or
4. the subjective experience of having alter personality self-states.
5. severe isolation of affect, with inability to feel body sensations or tune into emotions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Beck Scale for Suicide ideation (BSS) | Baseline
  21 item questionnaire on suicidal ideation and behaviour in past 1week. Score range 0 to 42, with higher scores worse in outcome.
Beck Scale for Suicide ideation (BSS) | 2 months after baseline
  21 item questionnaire on suicidal ideation and behaviour in past 1week. Score range 0 to 42, with higher scores worse in outcome.
Beck Scale for Suicide ideation (BSS) | 4 months after baseline
  21 item questionnaire on suicidal ideation and behaviour in past 1week. Score range 0 to 42, with higher scores worse in outcome.
Columbia Suicide Severity Rating Scale (CSSRS) Recent (self report of past 1 week) | Baseline
  6 questions on suicidal ideation. First Questions 3, 4, and 5 are answered only if Question 2 ("Have you actually had any thoughts of killing yourself") is answered as a yes. Questions 3 to 5 elaborate on suicidal ideation. Scored as "yes or no" for each question, as dichotomous variables.
Columbia Suicide Severity Rating Scale (CSSRS) Recent (self report of past 1 week) | 2 months
  6 questions on suicidal ideation. First Questions 3, 4, and 5 are answered only if Question 2 ("Have you actually had any thoughts of killing yourself") is answered as a yes. Questions 3 to 5 elaborate on suicidal ideation. Scored as "yes or no" for each question, as dichotomous variables.
Columbia Suicide Severity Rating Scale (CSSRS) Recent (self report of past 1 week) | 4 months
  6 questions on suicidal ideation. First Questions 3, 4, and 5 are answered only if Question 2 ("Have you actually had any thoughts of killing yourself") is answered as a yes. Questions 3 to 5 elaborate on suicidal ideation. Scored as "yes or no" for each question, as dichotomous variables.

SECONDARY OUTCOMES:
ACES Questionnaire (ACES) | Baseline only
  10 questions about childhood adversity, which can be added. Score ranges from 0 to 10, with higher number indicating worse adversity before age 18.
DES II (Dissociative Experiences Scale II). | Baseline
  28 item scale, with score ranging from 0 to 100, with higher score indicating higher dissociative symptoms and severity.
DES II (Dissociative Experiences Scale II). | 4 months after baseline
  28 item scale, with score ranging from 0 to 100, with higher score indicating higher dissociative symptoms and severity.
BDI II (Beck Depression Inventory II) | Baseline
  21 item questionnaire on depressive symptoms, score ranges from 0 to 63, with higher scores indicating worse depression.
BDI II (Beck Depression Inventory II) | 2 months after baseline
  21 item questionnaire on depressive symptoms, score ranges from 0 to 63, with higher scores indicating worse depression.
BDI II (Beck Depression Inventory II) | 4 months after baseline
  21 item questionnaire on depressive symptoms, score ranges from 0 to 63, with higher scores indicating worse depression.
PHQ-9 (Patient Health Questionnaire 9). | Baseline
  Nine item questionnaire on depressive symptoms, ranging from 0 (not at all) to 3 (nearly every day) for each item, scores range from 0 to 27 (worst symptoms). Then symptoms ranked as either Not difficult, somewhat difficult, Very difficult or Extremely difficult.
PHQ-9 (Patient Health Questionnaire 9). | 2 months after baseline
  Nine item questionnaire on depressive symptoms, ranging from 0 (not at all) to 3 (nearly every day) for each item, scores range from 0 to 27 (worst symptoms). Then symptoms ranked as either Not difficult, somewhat difficult, Very difficult or Extremely difficult.
PHQ-9 (Patient Health Questionnaire 9). | 4 months after baseline
  Nine item questionnaire on depressive symptoms, ranging from 0 (not at all) to 3 (nearly every day) for each item, scores range from 0 to 27 (worst symptoms). Then symptoms ranked as either Not difficult, somewhat difficult, Very difficult or Extremely difficult.
GAD 7 (Generalized Anxiety Disorder 7) | Baseline
  7 Item questionnaire on anxiety symptoms, each ranked from 0 (not at all) to 3 (nearly every day), with a score ranging from 0 to 21. Higher scores indicate worse anxiety.
GAD 7 (Generalized Anxiety Disorder 7) | 2 months after baseline
  7 Item questionnaire on anxiety symptoms, each ranked from 0 (not at all) to 3 (nearly every day), with a score ranging from 0 to 21. Higher scores indicate worse anxiety.
GAD 7 (Generalized Anxiety Disorder 7) | 4 months after baseline
  7 Item questionnaire on anxiety symptoms, each ranked from 0 (not at all) to 3 (nearly every day), with a score ranging from 0 to 21. Higher scores indicate worse anxiety.
IES-R (Impact of Events Revised) | Baseline
  22 item questionnaire on traumatic or stressful events. Each item ranges from 0 (not at all) to 4 (extremely), with scores ranging from 0 to 88 (higher is more severe).
IES-R (Impact of Events Revised) | 2 months after baseline
  22 item questionnaire on traumatic or stressful events. Each item ranges from 0 (not at all) to 4 (extremely), with scores ranging from 0 to 88 (higher is more severe).
IES-R (Impact of Events Revised) | 4 months after baseline
  22 item questionnaire on traumatic or stressful events. Each item ranges from 0 (not at all) to 4 (extremely), with scores ranging from 0 to 88 (higher is more severe).
DERS (Difficulties in Emotion Regulation Scale) | Baseline
  36 item questionnaire on emotion regulation, with each question ranked from 1 (almost never; 0-10% of the time) to 5 (almost always; 91-100% of the time). Scores range from 36 to 180, with higher scores indicating worse emotion regulation. Subscales indicate specific type of difficulties.
DERS (Difficulties in Emotion Regulation Scale) | 2 months after baseline
  36 item questionnaire on emotion regulation, with each question ranked from 1 (almost never; 0-10% of the time) to 5 (almost always; 91-100% of the time). Scores range from 36 to 180, with higher scores indicating worse emotion regulation. Subscales indicate specific type of difficulties.
DERS (Difficulties in Emotion Regulation Scale) | 4 months after baseline
  36 item questionnaire on emotion regulation, with each question ranked from 1 (almost never; 0-10% of the time) to 5 (almost always; 91-100% of the time). Scores range from 36 to 180, with higher scores indicating worse emotion regulation. Subscales indicate specific type of difficulties.
Healthcare care utilization | Comparing one year before to one year after study enrolment.
  Differences between the two arms with respect to number of emergency room visits and hospitalizations in the year before and after study.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Burback, MD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Hospital Edmonton - recruiting from AHS clinics internally, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
This is not in the plan.

REFERENCES:
- [Background] Fereidouni Z, Behnammoghadam M, Jahanfar A, Dehghan A. The Effect of Eye Movement Desensitization and Reprocessing (EMDR) on the severity of suicidal thoughts in patients with major depressive disorder: a randomized controlled trial. Neuropsychiatr Dis Treat. 2019 Aug 27;15:2459-2466. doi: 10.2147/NDT.S210757. eCollection 2019. PMID 31695382
- [Background] van Bentum JS, Sijbrandij M, Kerkhof AJFM, Huisman A, Arntz AR, Holmes EA, Franx G, Mokkenstorm J, Huibers MJH. Treating repetitive suicidal intrusions using eye movements: study protocol for a multicenter randomized clinical trial. BMC Psychiatry. 2019 May 9;19(1):143. doi: 10.1186/s12888-019-2129-0. PMID 31072317
- [Background] Bentum JSV, Sijbrandij M, Huibers MJH, Huisman A, Arntz A, Holmes EA, Kerkhof AJFM. Treatment of Intrusive Suicidal Imagery Using Eye Movements. Int J Environ Res Public Health. 2017 Jun 30;14(7):714. doi: 10.3390/ijerph14070714. PMID 28665329
- [Background] Van Woudenberg C, Voorendonk EM, Bongaerts H, Zoet HA, Verhagen M, Lee CW, van Minnen A, De Jongh A. Effectiveness of an intensive treatment programme combining prolonged exposure and eye movement desensitization and reprocessing for severe post-traumatic stress disorder. Eur J Psychotraumatol. 2018 Jul 10;9(1):1487225. doi: 10.1080/20008198.2018.1487225. eCollection 2018. PMID 30013726
- [Derived] Burback L, Yap S, Purdon SE, Abba-Aji A, O'Shea K, Bremault-Phillips S, Greenshaw AJ, Winkler O. Randomized controlled trial investigating web-based, therapist delivered eye movement desensitization and reprocessing for adults with suicidal ideation. Front Psychiatry. 2024 Feb 16;15:1361086. doi: 10.3389/fpsyt.2024.1361086. eCollection 2024. PMID 38435978
- [Derived] Winkler O, Dhaliwal R, Greenshaw A, O'Shea K, Abba-Aji A, Chima C, Purdon SE, Burback L. Web-Based Eye Movement Desensitization and Reprocessing for Adults With Suicidal Ideation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 4;10(11):e30711. doi: 10.2196/30711. PMID 34734835